CLINICAL TRIAL: NCT06109272
Title: A Phase 2/3, Randomized Study to Evaluate the Dose Optimization, Safety, and Efficacy of Livmoniplimab in Combination With Budigalimab in Subjects With Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) Who Have Not Previously Received Systemic Treatment
Brief Title: A Study to Assess the Dose, Adverse Events, and Change in Disease Activity of Livmoniplimab as an Intravenous (IV) Solution in Combination With Budigalimab as an IV Solution in Adult Participants With Hepatocellular Carcinoma (HCC)
Acronym: LIVIGNO-2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-052; 2023-504600-28-00 (Other: EU CT)
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Livmoniplimab; ABBV-151; budigalimab; ABBV-181
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — budigalimab; durvalumab; atezolizumab; Bevacizumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Stage 1: Cohort 1 (Experimental): Participants will receive livmoniplimab Dose 1 in combination with budigalimab every 3 weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Stage 1: Cohort 2 (Experimental): Participants will receive livmoniplimab Dose 2 in combination with budigalimab every 3 weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Stage 1: Cohort 3 - Group 1 (Control) (Active Comparator): Participants will receive atezolizumab in combination with bevacizumab every 3 weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Stage 1: Cohort 3 - Group 2 (Control) (Active Comparator): Participants will receive a single dose of tremelimumab in combination with durvalumab every four weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Stage 2: Arm 1 (Experimental): Participants will receive livmoniplimab (optimized dose) in combination with budigalimab every 3 weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Stage 2: Arm 2 (Control) (Active Comparator): Participants will receive a single dose of tremelimumab in combination with durvalumab every 4 weeks until disease progression or until discontinuation criteria are met.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Livmoniplimab — Intravenous (IV) Solution
  Other Names: ABBV-151
  Arms: Stage 1: Cohort 1; Stage 1: Cohort 2; Stage 2: Arm 1
Drug: Budigalimab — Intravenous (IV) Solution
  Other Names: ABBV-181
  Arms: Stage 1: Cohort 1; Stage 1: Cohort 2; Stage 2: Arm 1
Drug: Durvalumab — Intravenous (IV) Solution
  Arms: Stage 1: Cohort 3 - Group 2 (Control); Stage 2: Arm 2 (Control)
Drug: Atezolizumab — Intravenous (IV) Solution
  Arms: Stage 1: Cohort 3 - Group 1 (Control)
Drug: Bevacizumab — Intravenous (IV) Solution
  Arms: Stage 1: Cohort 3 - Group 1 (Control)
Drug: Tremelimumab — Intravenous (IV) Solution
  Arms: Stage 1: Cohort 3 - Group 2 (Control); Stage 2: Arm 2 (Control)

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cancer worldwide and a leading cause of cancer-related death. The majority of participants first presenting with HCC have advanced unresectable or metastatic disease. The purpose of this study is to evaluate the optimized dose, adverse events, and efficacy of livmoniplimab in combination with budigalimab.

Livmoniplimab is an investigational drug being developed for the treatment of HCC. There are 2 stages to this study. In Stage 1, there are 3 treatment arms and participants will be randomized in a 1:1:1 ratio. Participants will either receive livmoniplimab (at different doses) in combination with budigalimab (another investigational drug), atezolizumab in combination with bevacizumab, or tremelimumab in combination with durvalumab. In Stage 2, there are 2 treatments arms and participants will be randomized in a 1:1 ratio. Participants will either receive livmoniplimab (optimized dose) in combination with budigalimab or tremelimumab in combination with durvalumab. Approximately 660 adult participants will be enrolled in the study across 185 sites worldwide.

Stage 1: In arm 1, participants will receive intravenously (IV) infused livmoniplimab (Dose 1) in combination with IV infused budigalimab, every 3 weeks. In arm 2, participants will receive IV infused livmoniplimab (Dose 2) in combination with IV infused budigalimab, every 3 weeks. In Arm 3 (control), participants will receive the investigator's choice: IV atezolizumab in combination with IV bevacizumab every 3 weeks or single dose IV tremelimumab in combination with IV durvalumab every 4 weeks. Stage 2: In arm 1, participants will receive IV infused livmoniplimab (optimized dose) in combination with IV infused budigalimab, every 3 weeks. In Arm 2 (control), participants will receive single dose IV tremelimumab in combination with IV durvalumab every 4 weeks. All participants will continue treatment until disease progression or discontinuation criteria are met, whichever occurs first. The estimated duration of this study is about 56 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable hepatocellular carcinoma (HCC) with diagnosis confirmed by histology or cytology or clinically by American Association for the Study of Liver Diseases criteria for participants with cirrhosis.
* Barcelona Clinic Liver Cancer (BCLC) Stage B or C.
* Child-Pugh A or B7 classification (i.e., total Child-Pugh score of 5, 6, or 7).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.

Exclusion Criteria:

* Prior systemic therapy for HCC.
* Symptomatic, untreated, or actively progressing CNS metastases.
* History of malignancy other than HCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Best Overall Response (BOR) per Investigator | Through Study Completion, Up to Approximately 56 Months
  BOR is defined as a participant achieving confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by investigators at any time prior to subsequent anticancer therapy.
Stage 2: Overall Survival (OS) | Through Study Completion, Up to Approximately 56 Months
  OS is defined as the time from randomization until death from any cause

SECONDARY OUTCOMES:
Stage 1: Number of Participants with Progression-Free Survival (PFS) | Through Study Completion, Up to Approximately 56 Months
  PFS is defined as the time from randomization until the first documentation of progressive disease according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Stage 1: Duration of Response (DOR) per Investigator | Through Study Completion, Up to Approximately 56 Months
  DOR is defined as the time from first confirmed CR or PR until the first documentation of progressive disease according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Stage 1: Overall Survival (OS) | Through Study Completion, Up to Approximately 56 Months
  OS is defined as the time from randomization until death from any cause.
Stage 1: Number of Participants with Adverse Events (AEs) | Through Study Completion, Up to Approximately 56 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Stage 1: Maximum Plasma Concentration (Cmax) of Livmoniplimab and Budigalimab | Through Study Completion, Up to Approximately 56 Months
  Cmax of livmoniplimab and budigalimab.
Stage 1: Time to Cmax (Tmax) of Livmoniplimab and Budigalimab | Through Study Completion, Up to Approximately 56 Months
  Tmax of livmoniplimab and budigalimab.
Stage 1: Area Under the Serum Concentration Versus Time Curve (AUC) of Livmoniplimab and Budigalimab | Through Study Completion, Up to Approximately 56 Months
  AUC of livmoniplimab and budigalimab.
Stage 2: Number of Participants with Progression-Free Survival (PFS) | Through Study Completion, Up to Approximately 56 Months
  PFS is defined as the time from randomization until the first documentation of progressive disease according to RECIST 1.1 as determined blinded independent central review (BICR) or death from any cause, whichever occurs first.
Stage 2: Best Overall Response (BOR) of Complete Response (CR)/Partial Response (PR) per BICR | Through Study Completion, Up to Approximately 56 Months
  BOR is defined as a participant achieving confirmed CR/PR per RECIST 1.1 as determined by BICR at any time prior to subsequent anticancer therapy.
Change from Baseline in the Pain Domain of the European Organization for Research Treatment of Cancer Quality of Life Questionnaire Hepatocellular Carcinoma 18-Question Module (EORTC QLQ-HCC18) | Baseline to Week 12
  The EORTC QLQ-HCC18 is an 18-item scale that measures hepatocellular carcinoma (HCC)-specific symptoms and health-related quality of life (HRQoL). The Pain Domain contains 2 items where scores are based on a 4-point Likert scale (with 1 = 'not at all' to 4 = 'very much'); scaled scores for each domain ranged from 0-100 with a higher score indicating worse symptoms.
Change from Baseline in the Fatigue Domain of the EORTC QLQ-HCC18 | Baseline to Week 12
  The EORTC QLQ-HCC18 is an 18-item scale that measures HCC-specific symptoms and HRQoL. The Fatigue Domain contains 3 items where scores are based on a 4-point Likert scale (with 1 = 'not at all' to 4 = 'very much'); scaled scores for each domain ranged from 0-100 with a higher score indicating worse symptoms.
Change from Baseline in Physical Function (PF) Domain of the European Organization for Research Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) | Baseline to Week 12
  The EORTC QLQ-C30 is an 30-item patient-reported questionnaire that measures symptoms and HRQoL. The PF Domain is a functional scale where participants rate items on a 4-point scale (with 1 = 'not at all' to 4 = 'very much'). A change of 5 to 10 points is considered a small change and the lower bound (5) will be used to define the minimum important difference. A change of >= 10 to < 20 points is considered a moderate change.
Change from Baseline in Global Health Status (GHS)/Quality of Life (QoL) Domain as Measured by the GHS/QoL Domain of the EORTC QLQ-C30 | Baseline to Week 12
  The EORTC QLQ-C30 is an 30-item patient-reported questionnaire that measures symptoms and HRQoL. The GHS/QoL Domain is a scale where participants rate items on a 4-point scale (with 1 = 'not at all' to 4 = 'very much'). A change of 5 to 10 points is considered a small change and the lower bound (5) will be used to define the minimum important difference. A change of ≥ 10 to < 20 points is considered a moderate change.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (13):
  - City of Hope /ID# 261468, Duarte, California
  - City of Hope at Orange County Lennar Foundation Cancer Center /ID# 261669, Irvine, California
  - UC Irvine /ID# 255673, Orange, California
  - The University of Chicago Medical Center /ID# 255674, Chicago, Illinois
  - Alliance for Multispecialty Research LLC Kansas City Oncology /ID# 256830, Merriam, Kansas
  - Norton Cancer Institute /ID# 260775, Louisville, Kentucky
  - Henry Ford Hospital /ID# 255803, Detroit, Michigan
  - Metro Minnesota Community Oncology Research Consortium (MMCORC) /ID# 256041, Saint Louis Park, Minnesota
  - Washington University-School of Medicine /ID# 255720, St Louis, Missouri
  - Texas Oncology - Abilene - Antilley Road /ID# 265820, Abilene, Texas
  - Texas Oncology - Dallas - Worth Street /ID# 265806, Dallas, Texas
  - Baylor Scott and White Research Institute /ID# 260853, Dallas, Texas
  - Oncology and Hematology Associates of Southwest Virginia /ID# 265834, Roanoke, Virginia
- France (4):
  - CHU Grenoble - Hopital Michallon /ID# 256627, La Tronche, Isere
  - Institut Gustave Roussy /ID# 258460, Villejuif, Val-de-Marne
  - Hôpital Avicenne /ID# 266005, Bobigny, Île-de-France Region
  - Hopital Beaujon /ID# 256551, Clichy, Île-de-France Region
- Italy (7):
  - IRCCS Istituto Clinico Humanitas /ID# 256684, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 256404, Milan, Milano
  - P.O. Ospedale del Mare /ID# 256410, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 265506, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 256412, Bologna
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 256681, Palermo
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 256895, Roma
- Puerto Rico Medical Research Center /ID# 262362, Hato Rey, Puerto Rico, Puerto Rico
- Spain (7):
  - Hospital Universitario Marques de Valdecilla /ID# 255769, Santander, Cantabria
  - Hospital Universitario Reina Sofia /ID# 255779, Córdoba, Cordoba
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 255778, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron /ID# 255771, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 255772, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 255776, Seville
  - Hospital Universitario Miguel Servet /ID# 255774, Zaragoza
- Taiwan (5):
  - National Taiwan University Hospital /ID# 256168, Taipei City, Taipei
  - China Medical University Hospital /ID# 256764, Taichung
  - Taichung Veterans General Hospital /ID# 259405, Taichung
  - National Cheng Kung University Hospital /ID# 256766, Tainan
  - Taipei Veterans General Hosp /ID# 256169, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-052